CLINICAL TRIAL: NCT02562989
Title: A Study to Qualify [18F]MK-6240 Positron Emission Tomography (PET) for Use as a Biomarker of Neurofibrillary Tangle Pathology in Alzheimer's Disease
Brief Title: [18F]MK-6240 Positron Emission Tomography (PET) Tracer First-in-Human Validation Study (MK-6240-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 6240-001; 2015-001659-58 (EudraCT Number); MK-6240-001 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer's Disease; Amnestic Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1, Healthy Young Participants (Experimental): Healthy young participants received a single intravenous (IV) dose of ~185 megabecquerel (MBq) [18F]MK-6240 in Part 1 of the study
  Interventions: Drug: [18F]MK-6240, ~185 MBq
- Part 2, Healthy Elderly Participants (Experimental): Healthy elderly participants received a single IV dose of ~160 MBq [18F]MK-6240, in Part 2 of the study
  Interventions: Drug: [18F]MK-6240, ~160 MBq
- Part 2, AD and Amnestic MCI Elderly Participants (Experimental): AD and amnestic MCI participants received up to two IV doses of ~160 MBq [18F]MK-6240 in Part 2 of the study
  Interventions: Drug: [18F]MK-6240, ~160 MBq

INTERVENTIONS:
Drug: [18F]MK-6240, ~185 MBq — IV dose of ~185 MBq [18F]MK-6240
  Arms: Part 1, Healthy Young Participants
Drug: [18F]MK-6240, ~160 MBq — IV dose of ~160 MBq [18F]MK-6240
  Arms: Part 2, AD and Amnestic MCI Elderly Participants; Part 2, Healthy Elderly Participants

SUMMARY:
This 2-part, open-label study was designed to investigate the safety, tolerability, and efficacy of [18F]MK-6240, a Positron Emission Tomography (PET) imaging agent, for the quantification of neurofibrillary tangle (NFT) deposition in the brain. Brain NFT deposition is a pathologic finding in Alzheimer's Disease (AD), with brain NFT density shown to correlate with the severity of cognitive impairment in AD. The objectives of the study include performing the following with respect to [18F]MK-6240 administered as a PET imaging agent: 1) assess safety and tolerability; 2) determine radiation safety profile; 3) determine optimal imaging protocol parameters for quantification of brain NFTs in AD; 4) compare tracer binding in brain PET scans from participants with AD, participants with amnestic mild cognitive impairment (MCI) and healthy elderly participants; and 5) evaluate intra-subject test-retest (T-RT) variability of tracer uptake in brain regions of interest.

ELIGIBILITY:
Inclusion Criteria:

Part 1 and Part 2:

* Male, or non-pregnant and non-breast feeding female; in addition:

  * Male participant who is sexually active with females of childbearing potential must be willing to use a condom from the first dose of study drug until 3 months post the last dose of study drug
  * Female participant with reproductive potential must have serum β-human chorionic gonadotropin (β-hCG) test result consistent with non-pregnant state at screening and agree to use two acceptable methods of birth control beginning at screening visit, during study and until 2 weeks after the last dose of study drug
  * Post-menopausal female participant has been without menses for at least 1 year and has a documented follicle stimulating hormone (FSH) level in the postmenopausal range at screening
  * Surgically sterile female participant may enroll in study if procedure (hysterectomy, oophorectomy, or tubal ligation) is documented/confirmed by medical records or protocol-defined examination/tests
* Nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 3 months

Part 1 only:

* 18 to 55 years of age
* Body Mass Index (BMI) between 18-32 kg/m^2
* In good health based on medical history, physical examination, vital sign measurements, electrocardiogram (ECG) and laboratory safety tests

Part 2 only:

* 56 to 85 years of age
* Body weight <136 kg
* In stable medical condition based on medical history, physical examination, vital sign measurements and ECG
* In good health based on laboratory safety tests
* For some participants, willing to allow placement of an arterial catheter in the radial artery
* For AD participants:

  * Mini-Mental State Examination (MMSE) score ≤28
  * Meets National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for probable AD
  * Meets Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria for AD
  * Modified Hachinski score ≤4
  * Screening magnetic resonance imaging (MRI) scan consistent with a diagnosis of AD
  * Able to read at a 6th grade level or equivalent and has a history of academic achievement and/or employment sufficient to exclude mental retardation
  * Has a reliable informant/caregiver who is able to accompany the participant to all clinic visits and provide information to study investigator/staff via telephone contact
  * If taking symptomatic treatment for AD, be on a stable dose for at least 4 weeks prior to study
* For amnestic MCI participants:

  * MMSE score ≥26
  * A history of subjective memory decline before screening
  * Objective impairment in verbal memory based on investigator's clinical assessment
  * General cognitive function and activities of daily living sufficiently intact, so as not to meet criteria for mild AD dementia
  * Modified Hachinski score ≤4
  * MRI scan obtained at the screening visit is either normal or consistent with a diagnosis of AD
  * Able to read at a 6th grade level or equivalent and has a history of academic achievement and/or employment sufficient to exclude mental retardation
* For non-AD/non-MCI healthy elderly participants:

  * MMSE score ≥27
  * No history of subjective memory or other cognitive complaints
  * No objective evidence of memory or cognitive impairment

Exclusion Criteria:

Part 1 and Part 2:

* Subject has participated in another investigational trial within 4 weeks of screening
* Subject has participated in a PET research study or other study involving administration of a radioactive substance or ionizing radiation within 12 months prior to screening or has undergone an extensive radiological examination within this period
* History within 2 years prior to screening, or current evidence of a psychotic disorder or a major depressive disorder
* History of alcoholism or drug dependency/abuse within the last 2 years before screening
* History of cancer
* History of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Has positive test result for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* Participant has had major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to screening
* QTc interval ≥470 msec (for males) or ≥480 msec (for females)
* Participant consumes >3 servings of alcohol a day
* Participant consumes >6 caffeine servings a day
* Participant is currently a regular or recreational user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 3 months
* Suffers from claustrophobia or an inability to tolerate confinement in small places and would be unable to undergo PET or (for Part 2 only) MRI scanning

Part 1 Only:

* Evidence of a clinically relevant neurological disorder at screening
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological abnormality or disease
* Participant is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies, beginning approximately 2 weeks prior to administration of the initial dose of study drug and throughout the study

Part 2 Only:

* Evidence of a clinically relevant neurological disorder other than AD at screening
* History or current evidence of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological abnormality or disease, which is not adequately controlled through a stable medication regimen
* Participant has or is suspected to have implanted or embedded metal objects, or fragments in the head or body that would present a risk during the MRI scanning procedure
* For participants undergoing arterial catheter placement only:

  * Allergy to lidocaine which may be locally injected as an anesthetic
  * Currently uses aspirin or aspirin-containing medications at doses exceeding 100 mg daily, or nonsteroidal anti-inflammatory drugs (NSAIDs), which cannot be discontinued 2 weeks prior to dosing and throughout the course of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2016-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lohith TG, Bennacef I, Vandenberghe R, Vandenbulcke M, Salinas CA, Declercq R, Reynders T, Telan-Choing NF, Riffel K, Celen S, Serdons K, Bormans G, Tsai K, Walji A, Hostetler ED, Evelhoch JL, Van Laere K, Forman M, Stoch A, Sur C, Struyk A. Brain Imaging of Alzheimer Dementia Patients and Elderly Controls with 18F-MK-6240, a PET Tracer Targeting Neurofibrillary Tangles. J Nucl Med. 2019 Jan;60(1):107-114. doi: 10.2967/jnumed.118.208215. Epub 2018 Jun 7. PMID 29880509

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 2, AD and Amnestic MCI Elderly Participants: AD and amnestic MCI participants received up to two IV doses of ~160 MBq [18F]MK-6240, in Part 2 of the study.
Period: Overall Study
Arm/Group | Part 1, Healthy Young Participants | Part 2, Healthy Elderly Participants | Part 2, AD and Amnestic MCI Elderly Participants
Started | 3 | 4 | 6
Completed | 3 | 4 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Healthy Young Participants | Part 2, Healthy Elderly Participants | Part 2, AD and Amnestic MCI Elderly Participants | Total
Number analyzed (Participants) | 3 | 4 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.0 (7.9) | 65.3 (5.4) | 73.2 (4.4) | 60.1 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 1 | 3 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: The number of participants experiencing an adverse event (AE) was monitored. An AE is any unfavorable and unintended medical occurrence, symptom, or disease witnessed in a participant, regardless of whether or not a causal relationship with the study treatment can be demonstrated. Further, any worsening of a preexisting condition that is temporally associated with the use of the study treatment is also considered an AE.
Time Frame: Part 1: Up to 5 weeks; Part 2: up to 16 weeks
Population: All participants as treated, consisting of all participants who received at least 1 dose of [18F]MK-6240
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Healthy Young Participants | Part 2, Healthy Elderly Participants | Part 2, AD and Amnestic MCI Elderly Participants
Number analyzed (Participants) | 3 | 4 | 6
Participants | 1 | 3 | 2

2. Primary Outcome: Number of Participants Who Discontinued Study Due to an AE
Description: The number of participants discontinuing study due to an AE was monitored.
Time Frame: Part 1: Up to 5 weeks; Part 2: up to 16 weeks
Population: All participants as treated, consisting of all participants who received at least 1 dose of [18F]MK-6240
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Healthy Young Participants | Part 2, Healthy Elderly Participants | Part 2, AD and Amnestic MCI Elderly Participants
Number analyzed (Participants) | 3 | 4 | 6
Participants | 0 | 0 | 0

3. Primary Outcome: Effective Dose of [18F]MK-6240
Description: Mean effective dose (ED) of [18F]MK-6240 was calculated from whole-body (WB) PET scans of healthy young participants included in Part 1 of study. ED, reported as microsieverts (µSv) / megabecquerel (MBq), is a measure of WB radiation exposure risk that accounts for differences in individual organ exposure and organ susceptibility to ionizing radiation. Following [18F]MK-6240 PET tracer administration, organ-specific time-activity curves (TACs) and radioactivity residence times were utilized to calculate exposure risk for individual organs. These values calculated for individual organs were then entered into a human biodistribution model to determine ED of [18F]MK-6240.
Time Frame: Up to approximately 5 hours following [18F]MK-6240 administration
Population: The analysis population included only healthy young participants enrolled in Part 1 of this study (N=3). As per study protocol, participants enrolled in Part 2 did not receive testing for effective dose of [18F]MK-6240 and, as a result, were not included in the analysis population.
Measure: Mean (Standard Deviation); unit: µSv / MBq
Arm/Group | Part 1, Healthy Young Participants | Part 2, Healthy Elderly Participants | Part 2, AD and Amnestic MCI Elderly Participants
Number analyzed (Participants) | 3 | 0 | 0
µSv / MBq | 29.4 (0.6) |  |

4. Primary Outcome: Organ Effective Dose of [18F]MK-6240
Description: Mean organ ED of [18F]MK-6240 was calculated from WB PET scans of healthy young participants included in Part 1 of study. Organ ED, reported as micrograys (µGy) / MBq, is a measure of organ-specific radiation exposure risk. Following [18F]MK-6240 PET tracer administration, organ-specific TACs and radioactivity residence times were utilized to calculate organ ED for specific organs of the body.
Time Frame: Up to approximately 5 hours following [18F]MK-6240 administration
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µGy / MBq
Arm/Group | Part 1, Healthy Young Participants | Part 2, Healthy Elderly Participants | Part 2, AD and Amnestic MCI Elderly Participants
Number analyzed (Participants) | 3 | 0 | 0
µGy / MBq
  Adrenals | 12.7 (1.0) |  |
  Brain | 8.8 (0.4) |  |
  Breasts | 5.8 (0.9) |  |
  Gallbladder Wall | 202.0 (111.0) |  |
  Lower Large Intestine Wall | 46.4 (5.5) |  |
  Small Intestine | 116.0 (13.3) |  |
  Stomach Wall | 16.9 (3.7) |  |
  Upper Large Intestine Wall | 128.0 (15.7) |  |
  Heart Wall | 15.6 (1.0) |  |
  Kidneys | 33.5 (4.8) |  |
  Liver | 34.3 (9.2) |  |
  Lungs | 19.7 (3.6) |  |
  Muscle | 9.4 (0.8) |  |
  Ovaries | 28.3 (2.0) |  |
  Pancreas | 14.6 (1.1) |  |
  Red Marrow | 19.2 (2.9) |  |
  Osteogenic Cells | 16.9 (1.5) |  |
  Skin | 5.6 (0.8) |  |
  Spleen | 17.7 (3.9) |  |
  Testes | 3.0 (5.1) |  |
  Thymus | 6.9 (1.1) |  |
  Thyroid | 5.6 (1.5) |  |
  Urinary Bladder Wall | 128.0 (31.8) |  |
  Uterus | 26.4 (1.2) |  |

5. Primary Outcome: Standardized Uptake Value Ratio (SUVR) of [18F]MK-6240 in Brain Regions of Interest
Description: As a surrogate of regional [18F[MK-6240 tracer distribution volume (VT), mean standardized uptake value ratios (SUVRs), were calculated for specific brain regions of interest (ROIs) in healthy elderly as well as AD/MCI elderly participants in Part 2 of the study. Calculated using calibrated PET scan images from each participant, SUVR is the relative ratio of pixel intensities at a specific brain ROI compared to a reference region (RR; cerebellar cortex, for this study). For an individual participant, the average SUVR for each brain ROI is calculated starting at 60 minutes and ending at 90 minutes following [18F]MK-6240 administration to quantify tracer retention; referred to as "SUVR (60-90min)."
  An SUVR (60-90 min) < 1 indicates decreased tracer retention at brain ROI relative to RR.
  An SUVR (60-90 min) = 1 indicates no difference in tracer retention at brain ROI relative to RR.
  An SUVR (60-90 min) > 1 indicates increased tracer retention at brain ROI relative to RR.
Time Frame: From 60 to 90 minutes following [18F]MK-6240 administration
Population: The analysis population included healthy elderly as well as AD/amnesic MCI participants enrolled in Part 2 of this study. As per study protocol, participants enrolled in Part 1 did not receive testing for SUVR (60-90 min) and, as a result, were not included in the analysis population.
Measure: Mean (Standard Deviation); unit: SUVR (60-90 min)
Arm/Group | Part 1, Healthy Young Participants | Part 2, Healthy Elderly Participants | Part 2, AD and Amnestic MCI Elderly Participants
Number analyzed (Participants) | 0 | 4 | 6
SUVR (60-90 min)
  Frontal Lobe |  | 0.95 (0.07) | 1.22 (0.47)
  Temporal Lobe |  | 0.98 (0.07) | 1.64 (0.72)
  Parietal Lobe |  | 0.95 (0.06) | 1.42 (0.80)
  Occipital Lobe |  | 1.01 (0.06) | 1.61 (0.92)
  Insula and Cingulate Cortex |  | 0.93 (0.07) | 1.22 (0.42)
  Hippocampus |  | 0.93 (0.10) | 1.37 (0.25)
  Amygdala |  | 0.84 (0.11) | 1.67 (0.40)
  Parahippocampal and Ambient Gyri |  | 0.96 (0.11) | 1.71 (0.39)
  Fusiform Gyri |  | 1.03 (0.11) | 1.72 (0.67)
  Striatum |  | 0.86 (0.04) | 0.92 (0.21)
  Thalamus |  | 0.85 (0.06) | 0.81 (0.13)
  Substantia Nigra |  | 1.10 (0.11) | 1.08 (0.14)
  Brainstem |  | 0.78 (0.09) | 0.76 (0.09)

6. Primary Outcome: Intra-subject Test-Retest (T-RT) Variability of Standardized Uptake Value Ratio (SUVR) in Brain Regions of Interest
Description: For each AD/MCI participant receiving 2 doses of MK-6240, the SUVR (60-90 min) during initial dose (SUVR_1) was compared to the SUVR (60-90 min) during the second dose (SUVR_2) to determine the percent test-retest (T-RT) variability of the SUVR (60-90 min) for each brain ROI.
  T-RT variability = (absolute value (SUVR_1 - SUVR_2) / average SUVR) * 100. If T-RT variability = 0, indicates no variability between SUVR_1 and SUVR_2.
Time Frame: Up to 16 weeks following initial dose of [18F]MK-6240
Population: Includes only elderly AD/MCI participants (Part 2); per protocol, young (Part 1) and elderly (Part 2) healthy participants did not receive retest scan. Of the 6 AD/MCI participants, only 2 received T-RT scans. In one participant, motion artifacts prevented T-RT analysis. For the one participant included, T-RT scans were separated by 16 weeks.
Measure: Number; unit: Percent
Arm/Group | Part 1, Healthy Young Participants | Part 2, Healthy Elderly Participants | Part 2, AD and Amnestic MCI Elderly Participants
Number analyzed (Participants) | 0 | 0 | 1
Percent
  Frontal Lobe |  |  | 7
  Temporal Lobe |  |  | 12
  Parietal Lobe |  |  | 7
  Occipital Lobe |  |  | 9
  Insula and Cingulate Cortex |  |  | 4
  Hippocampus |  |  | 6
  Amygdala |  |  | 5
  Parahippocampal and Ambient Gyri |  |  | 6
  Fusiform Gyri |  |  | 17
  Striatum |  |  | 4
  Thalamus |  |  | 2
  Substantia Nigra |  |  | 6
  Brainstem |  |  | 2

ADVERSE EVENTS:
Time Frame: Part 1: up to 5 weeks Part 2: up to 16 weeks
Arm/Group | Part 1, Healthy Young Participants | Part 2, Healthy Elderly Participants | Part 2, AD and Amnestic MCI Elderly Participants
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 1/3 | 3/4 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Healthy Young Participants (N=3) | Part 2, Healthy Elderly Participants (N=4) | Part 2, AD and Amnestic MCI Elderly Participants (N=6)
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Vascular access site hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.